CLINICAL TRIAL: NCT02789488
Title: Efficacy and Safety of Furocyst in Patients With Poly Cystic Ovary Syndrome
Brief Title: Clinical Evaluation of Furocyst in Patients With Poly Cystic Ovary Syndrome
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chemical Resources (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CR001/PCOS-5-13
Record Dates: First submitted 2016-04-20; First posted 2016-06-03 (Estimated); Last update posted 2016-06-03 (Estimated); Status verified 2013-09

CONDITIONS: Poly Cystic Ovary Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Furocyst (Other): Furocyst one caps BID
  Interventions: Dietary Supplement: Fenugreek seeds extract 500 mg

INTERVENTIONS:
Dietary Supplement: Fenugreek seeds extract 500 mg — Furocyst one caps BID
  Other Names: Furocyst

SUMMARY:
Poly cystic ovary syndrome (PCOS) is a disease which is prevalent in women of reproductive age facing obesity along with increased risk of type-2 diabetes and high cholesterol levels. The genetically determined cause of the PCOS includes disturbed levels of insulin and androgens. Standardized fenugreek seed extract (Furocyst) contains compounds such as saponins & flavonoids which act on the insulin and indirectly helps to regulate the androgen levels in the body.

DETAILED DESCRIPTION:
Polycystic ovary syndrome is considered as clinical and public health consequence involving increase in number of cysts in women at reproductive age. These cysts are under-developed sacs in which eggs are developed. In PCOS, these sacs are unable to release an egg which means ovulation doesn't take place.

The estimated 5-10% prevalence of PCOS is reported in women of reproductive age. A study from Spain also reported that 28.3% prevalence rate of PCOS is among 113 overweight or obese women who were referred to an endocrinology clinic for weight loss. This data was compared with a previously reported prevalence of 6.5% which suggests that the prevalence of PCOS might be markedly increasing with obesity.

PCOS impacts significantly on various hormonal cycles. With PCOS, luteinizing hormone (LH) levels become higher than follicle stimulating hormone (FSH) levels. Because of this increase in LH levels, the LH surge does not take place and ovulation doesn't carry out which results in irregular menstrual cycle. The irregular menstrual period produces oligomenorrhea (few menstrual periods) or amenorrhea (no menstrual periods) and infertility due to irregular or lack of ovulation. PCOS also produces high levels of masculinizing hormones with symptoms of acne and hirsutism, hypermenorrhea involving heavy and prolonged menstrual periods and androgenic alopecia (increase hair thinning and diffused hair loss). The other metabolic syndromes associated with PCOS are increased risk of type 2 diabetes, high cholesterol levels and obesity.

These complications arise because of the genetically determined cause of the PCOS i.e. hyper- secretion of androgens from the ovary which favours excess luteinizing hormone (LH) secretion and insulin resistance. However, insulin resistance with or without a genetic mutation may be the initiator, followed by hyper-androgenism. Thus, insulin resistance is an important contributing factor to abnormal steroidogenesis in PCOS because hyper-insulinemia stimulates the pathway of insulin like growth factor-I (IGF-I) in theca cells of the ovary by cross-reacting with the receptors of IGF. Stimulation of the ovarian theca cells increases the production of androgens (eg, testosterone, androstenedione) which in turn, blocks the down-regulation of androgens by LH surge and leads to the hyper-androgenic environment in the ovary. Because of a decreased level of FSH relative to LH, the ovarian granulosa cells cannot aromatize the androgens to estrogens, which lead to decreased estrogen levels and results in anovulation.

Treatments for PCOS are chosen based on woman's symptoms, age and future pregnancy plans which may include birth control pills to regulate menstruation, insulin-sensitizing medications, ovulation induction to treat infertility, androgen-blocking medications, topical anti-hair-growth medications, etc.

Standardized fenugreek (Trigonella foenum graecum) seed extract (Furocyst) plays an important role in the management of PCOS. It improves glucose-tolerance and insulin-sensitivity, thereby promoting weight loss and moderation of androgen levels in the blood. Standardized fenugreek seeds extract contains a group of furostanolic saponins, derived from fenugreek seeds by an innovative process. It contains rich variety of saponins and flavonoids which have been known to lower the blood lipid levels and play valuable role in improving insulin sensitivity. Standardized fenugreek seeds extract is a dual insulin-sensitizer. In the presence of high fiber furostanolic saponins, cells become more sensitive to insulin & an increase in number of insulin receptor sites occurs. These receptor sites are responsive to insulin to stimulate the cells ability to burn glucose. This decrease in insulin resistance helps in the management of PCOS.

Considering the beneficial effects of standardized fenugreek seed extract, present study was conducted to evaluate the efficacy of fenugreek seeds extract in patients with poly cystic ovary syndrome by assessing reduction in ovarian volume and decrease in the number of ovarian cysts.

ELIGIBILITY:
Inclusion Criteria:

* Premenopausal women between 18-45 years of age and BMI less than 42
* Diagnosed with PCOS
* Adequate hepatic, renal and hematological functions
* Patients willing to give informed consent in writing

Exclusion Criteria:

* Males
* Post menopausal women
* Women with hysterectomy
* Patients with congenital adrenal hyperplasia
* Patients suffering from Cushing's syndrome
* Patients diagnosed with androgen secreting tumors
* Patients with thyroid dysfunction (T3, T4 level is higher than that in normal women of reproductive age)
* Patients with Hypo-gonadotropic and Hypo-gonadism (central origin of ovarian dysfunction)
* Pregnancy or desire for pregnancy or lactating mothers

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2013-09; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Reduction in Ovary volume as assessed by ultrasound | 12 weeks
  volume in cubic cms

CONTACTS AND LOCATIONS:
Overall Officials: Dr Amrita Sarkari Jaipuriar, MS, Principal Investigator — Garg Hospital,Goalghar .Gorakhpur,UP,India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ehrmann DA. Polycystic ovary syndrome. N Engl J Med. 2005 Mar 24;352(12):1223-36. doi: 10.1056/NEJMra041536. No abstract available. PMID 15788499
- [Background] Schroder AK, Tauchert S, Ortmann O, Diedrich K, Weiss JM. [Insulin resistance in polycystic ovary syndrome]. Wien Klin Wochenschr. 2003 Dec 15;115(23):812-21. doi: 10.1007/BF03041041. German. PMID 14740344
- [Background] Hassanzadeh Bashtian M, Emami SA, Mousavifar N, Esmaily HA, Mahmoudi M, Mohammad Poor AH. Evaluation of Fenugreek (Trigonella foenum-graceum L.), Effects Seeds Extract on Insulin Resistance in Women with Polycystic Ovarian Syndrome. Iran J Pharm Res. 2013 Spring;12(2):475-81. PMID 24250624